CLINICAL TRIAL: NCT01989949
Title: Phase 1, Open-Label, Safety and Pharmacokinetic Study to Assess Bronchopulmonary Disposition of Intravenous TP-434 in Healthy Men and Women
Brief Title: Safety and Pharmacokinetic (PK) Study to Assess Bronchopulmonary Disposition of IV Eravacycline (TP-434) in Healthy Men and Women
Acronym: BAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TP-434-006
Record Dates: First submitted 2013-09-10; First posted 2013-11-21 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Normal Drug Tolerance
MeSH Terms: interventions — eravacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TP-434 (Eravacycline) via IV infusion (Experimental): TP-434 (Eravacycline) reconstituted and administered via IV infusion at a dose of 1 mg/kg, every 12 hours, for 7 doses over 4 days.
  Interventions: Drug: TP-434 (Eravacycline) reconstituted and administered via an IV infusion

INTERVENTIONS:
Drug: TP-434 (Eravacycline) reconstituted and administered via an IV infusion

SUMMARY:
This is a phase 1, open-label, randomized pharmacokinetic and safety study in healthy adult subjects, who will undergo bronchoscopy and bronchoalveolar lavage (BAL) after receiving seven (7) doses of 1.0 mg/kg IV TP-434.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized pharmacokinetic and safety study in healthy adult subjects, who will undergo bronchoscopy and bronchoalveolar lavage (BAL) after receiving seven (7) doses of 1.0 mg/kg IV TP-434. Dosing will be twice daily (q12h) for three consecutive days beginning on day one (1) and a morning dose on day four (4).

Approximately 20 subjects will be enrolled into the study at one (1) investigational site. The population for this study is healthy male and female subjects 18 to 65 years of age.

This study includes a Screening Period of up to 30 days, a 4 day, open-label Treatment Period, and a two week Follow-up Period. There will be one 6 day/5 night inpatient stay (Days -1 to 5) during the Treatment Period and one outpatient visit at the end of the Follow-up Period. Excluding the Screening Period, the total duration of confinement (in the Clinical Research Center) will be approximately six (6) days and the total study duration, not including screening, will be approximately three (3) weeks.

Participants will be admitted to the Clinical Research Center on Day -1. Participants will receive four (4) days of intravenous TP-434 1.0 mg/kg of body weight twice daily (q12h) for three consecutive days and a morning dose on day four (4) (for a total of 7 doses) starting on Day 1. Blood and urine samples, ECGs, and vital signs will be collected for safety analysis at specified time points.

Pharmacokinetic blood sampling will occur on Day 4before and after the Day 4 dose of TP-434 at specified time points.

Participants will be randomized to a single BAL procedure time point. Bronchoscopy and BAL will be performed at the following time points after dosing of TP-434 on Day 4: two (2), four (4), six (6), and 12 hours after start of infusion. Bronchoscopy and BAL will be conducted for up to five (5) different participants at each time point. Each subject will undergo bronchoscopy and BAL only once.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age >18 to ≤ 65 years of age, inclusive
3. Body mass index of 18 to 33 kg/m2 or, if outside the range, considered not clinically significant by the Investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use adequate methods of contraception

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Subjects who have previously received TP-434
3. History of any drug or alcohol abuse in the past 2 years
4. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
5. Current smokers and those who have smoked within the last 6 months.
6. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator at screening
7. Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis as judged by the Investigator
8. Positive tests for drugs of abuse
9. Positive hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV; I and II) results
10. History of chronic respiratory disorders as judged by the Investigator
11. Serious adverse reaction or serious hypersensitivity to tetracyclines, midazolam or like compound, lidocaine or like compounds, or the formulation excipients
12. Donation or loss of greater than 400 mL of blood within the previous 3 months
13. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (with the exception of anti inflammatory, anti-hypertensive medications, or hormone replacement therapy) in the 14 days before Investigational Medicinal Product administration unless judged to not interfere with the study objectives according to the Investigator and sponsor's medical monitor
14. Failure to satisfy the Investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To determine the steady-state plasma pharmacokinetics and disposition of TP-434 into the epithelial lining fluid (ELF) and alveolar macrophages (AM) of healthy adult subjects after intravenous (IV) administration. | End of Therapy (Day 4)

SECONDARY OUTCOMES:
To determine the safety and tolerability of TP-434 in healthy adult subjects based primarily on the incidence, intensity and type of adverse events (AEs), clinical laboratory assessments, physical examinations, vital signs, and 12-lead ECGs. | Screening Visit through Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Horn, MD, PhD, Study Director — Tetraphase Pharmaceuticals, Inc
Locations (1):
- Center for Anti-infective Research and Development; Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Ji X-w, Mak WY, Xue F, Yang W-y, Kuan IH-S, Xiang X-q, Li Y, Zhu X. Population pharmacokinetics and pulmonary modeling of eravacycline and the determination of microbiological breakpoint and cutoff of PK/PD. Antimicrob Agents Chemother. 2025 Mar 5;69(3):e0106524. doi: 10.1128/aac.01065-24. Epub 2025 Jan 29. PMID 39878492